CLINICAL TRIAL: NCT02577068
Title: Combination Effect of Nefopam With Propacetamol for Postoperative Pain After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2015-0746
Record Dates: First submitted 2015-10-06; First posted 2015-10-16 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-02

CONDITIONS: Thyroidectomy; Pain
MeSH Terms: conditions — Pain | interventions — Nefopam; propacetamol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- nefopam group (Active Comparator)
  Interventions: Drug: Nefopam
- propacetamol group (Active Comparator)
  Interventions: Drug: Propacetamol
- nefopam and propacetamol group (Experimental)
  Interventions: Drug: Nefopam; Drug: Propacetamol

INTERVENTIONS:
Drug: Nefopam — Patients undergoing thyroidectomy receive medications depending on the group allocation 30minutes prior to the surgery end; Nefopam 20mg, Propacetamol 2g, and Nefopam 20mg+Propacetamol 2g. In addition, patients will take the same medication every six hours during POD 1.
  Arms: nefopam and propacetamol group; nefopam group
Drug: Propacetamol — Patients undergoing thyroidectomy receive medications depending on the group allocation 30minutes prior to the surgery end; Nefopam 20mg, Propacetamol 2g, and Nefopam 20mg+Propacetamol 2g. In addition, patients will take the same medication every six hours during POD 1.
  Arms: nefopam and propacetamol group; propacetamol group

SUMMARY:
Patients undergoing thyroidectomy are suffering not only surgical wound pain but posterior neck pain because of neck extension position during the surgery. However, there has been little attention of posterior neck pain. Nefopam and Propacetamol have different pharmacodynamics and been used for postoperative pain control in thyroidectomy patients. The aim of this study is evaluation of combination effect of Nefopam and Propacetamol for acute wound pain, posterior neck pain and chronic pain after thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* patient who undergone open thyroidectomy
* 20~70 years old
* ASA I~III

Exclusion Criteria:

* hypersensitivity on Nefopam and Propacetamol
* Liver failure, chronic alcohol addiction
* severe hemolytic anemia, chronic nutrition deficiency
* history of seizure
* MI, MAO inhibitor
* pregnant, breast-feeding
* foreigners

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-11-15; Primary Completion 2016-08-23 (Actual); Study Completion 2016-08-23 (Actual)

PRIMARY OUTCOMES:
VAS score on wound site and posterior neck | one hour after the surgery
  Patients' subject pain score through VAS on the surgery wound site and posterior neck.

SECONDARY OUTCOMES:
Additional pain rescue drug | for postop. 24hrs.
  how much of pain rescue drugs taken besides PCA
Postoperative nausea and vomiting | for postop. 24hrs.
  nausea score (0-none, 1- a little, 2- moderate, 3-severe) and vomiting (all or none)
Patient satisfaction | for postop. 24hrs.
  Patients satisfaction score ( 0- dissatisfaction, 1- a little dissatisfaction, 2- average, 3- a little satisfaction, 4- satisfaction)
Chronic pain and neurogenic pain | three month after the surgery.
  Neuropathic pain diagnostic questionnaire(DN 4) :
  The DN4 questionnaire consists of a total of 10 items grouped in 4 sections. The first seven items are related to the quality of pain (burning, painful cold, electric shocks) and its association to abnormal sensations (tingling, pins and needles, numbness, itching). The other 3 items are related to neurological examination in the painful area (touch hypoesthesia, pinprick hypoesthesia, tactile allodynia). A score of 1 is given to each positive item and a score of 0 to each negative item. The total score is calculated as the sum of all 10 items, and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10. All questions are related to pain which is the claim for current medical consultation.
acute VAS on wound site and posterior neck | postop. 24hrs.
  VAS for patients' subject pain scor

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Han DW, Koo BN, Chung WY, Park CS, Kim SY, Palmer PP, Kim KJ. Preoperative greater occipital nerve block in total thyroidectomy patients can reduce postoperative occipital headache and posterior neck pain. Thyroid. 2006 Jun;16(6):599-603. doi: 10.1089/thy.2006.16.599. PMID 16839262